CLINICAL TRIAL: NCT05536375
Title: A Pilot Feasibility Study of Detection of IL-11 and Other Cytokines in the Exhaled Breath Condensate (EBC) and Blood of Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022/2149
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 25 healthy adult volunteers who are:-
  1. Aged 21-65 years old with no pre-existing medical condition
  2. Not on any long term medication
  3. Non smoker
Masking Description: Participant will be assigned a research ID which will be used for sample and data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy volunteers (Other)
  Interventions: Other: Exhaled breath condensate collection and blood draw

INTERVENTIONS:
Other: Exhaled breath condensate collection and blood draw — Venepuncture- 10mls of blood to be collected
  and
  Exhaled breath condensate (EBC) collection method- this involved breathing in and out through a disposable device (akin to breathing onto cold glass to produce condensate) with an external cooler device. The R Tube starter kit is a complete disposable EBC collection kit and It has been used in many research clinical investigations.

SUMMARY:
IL-11 is a receptor previously proven to be highly expressed in human lungs with idiopathic lung fibrosis, and in animal model, IL-11 receptor neutralizing antibody has been shown to prevent the process of fibrosis in bleomycin-induced lung fibrosis in rats. Separately, investigators know the expression of IL-11 can be detected in human by measuring its expression in the exhaled breath condensate (EBC) and serum. With the sera obtained, investigators will examine a whole range of other interleukins which had been implicated in mammalian lung fibrosis.

Investigators aim to measure IL-11 in a pilot of human volunteers (healthy). This is important to subsequently see if IL-11 expression is increased in patients with a range of fibrotic diseases, with the potential to be used as diagnostic tool as well and to select patients who may benefit from IL-11 neutralizing antibody to delay/ cure their lung fibrosis including patients with idiopathic pulmonary fibrosis (IPF), drug/ radiation induced fibrosis and possibly even lung fibrosis as a chronic sequelae of COVID infection. IL-11 also has been shown to be highly relevant in cardiac patients- including chronic heart failure patients. Having reference ranges for IL-11 in the blood and EBC of healthy human volunteers will also be useful in future drug trials for IL-11 antibodies for future cardiac studies.

DETAILED DESCRIPTION:
IL-11 has been proven to be highly expressed in lungs of patients with idiopathic pulmonary fibrosis (IPF), a type of interstitial lung disease (ILD). An IL-11 neutralizing antibody has been shown to diminish lung inflammation and fibrosis in bleomycin induced lung fibrosis in mice model. In this study, IL-11 has also been shown to be expressed in samples of human lungs with IPF. The mechanism had been shown to be linked to reduction of fibroblast proliferation and activity.

The identification of individuals with different sub-types of lung fibrosis can be based on symptoms, lung function tests, radiology or even lung biopsies. However, all these methods are rather subjective and sometimes invasive but yet inconclusive. So to identify individual patients whom IL-11 may play a role in their disease processes, investigators propose to use IL-11 in EBC as a biomarker to identify these patients.

The design of this pilot study is; prospective, single arm, non-interventional study involving invasive investigations

1. Procedures/ investigations
2. Blood taking (venepuncture)
3. Exhaled breath condensate (EBC) collection method- this involved breathing in and out through a disposable device (akin to breathing onto cold glass to produce condensate) with an external cooler device. The R Tube starter kit is a complete disposable EBC collection kit that is FDA approved in USA. It has been used in many research clinical investigations. Investigators prefer completely disposable kits (not just mouthpiece).

Laboratory method in detection and quantification of IL-11 (ELISA)- Investigators will use the Human IL-11 Quantikine ELISA kit (#D1100, R&D Systems) to measure IL-11 concentrations in serum/ plasma, and EBC. This immunoassay has been used by Prof Cook's team for accurate quantification of IL-11 concentrations within the assay ranges of 31.2 - 2,000 pg/mL in studies, and possess a similar a detection range to that of another IL-11 ELISA kit used in a prior publication which quantified IL-11 concentrations in the serum and EBC. Each ELISA kit allows for simultaneous detection in up to 96 samples (including duplicates and standards). The assay employs the quantitative sandwich ELISA technique. Investigators may also use similar technique to examine the whole range of other interleukins which involved in lung fibrosis.

The use of EBC to detect IL-11 has been previously shown to be feasible and detectable in healthy volunteers. In that series, it was demonstrated that IL-11 levels were significantly increased in patients with NSCLC. Investigators first need to reproduce the feasibility of detection of IL-11 in EBC of healthy volunteers and use this as a reference range for levels of IL-11 in EBC of patients with fibrosis. IL-11 has previously been shown to be detectable in serum of human patients with pancreatitis by ELISA kits too. If this is the case, investigators can propose to use IL-11 as a screening tool, to identify patients who may benefit from IL-11 neutralizing antibody when this is available in humans.

Other interleukins which have been shown to contribute to lung fibrosis are IL-1B and IL-5, in rat animal models, by promoting inflammation. IL-9, IL-10, and IL-17 on the other hand are protective in lung fibrosis. IL-12 inhibits collagen synthesis. IL-2, IL-4, IL-6, IL-13, IL-18 and IL-37 have also been shown to contribute to lung fibrosis through cell proliferation and fibroblasts activation, rather than direct inflammation. More importantly, IL-2, IL-6, IL-8, IL-10, and IL-12 have been shown to be increased in sera of patients with IPF compared to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21-65 years old with no pre-existing medical condition
2. Not on any long term medication
3. Non smoker

Exclusion Criteria:

1. Previous myocardial infarction (MI), inclusive of ST-elevation MI (STEMI) and non-ST-elevation MI (NSTEMI)
2. Known coronary artery disease or known flow limiting CAD (>75% stenosis)
3. Prior cardiac surgery (including but not limited to PCI, CABG, ICD/PPM implant etc)
4. BMI>35
5. Alcohol intake >10 units per week
6. Known definite diabetes mellitus or on treatment for diabetes mellitus
7. Asthma or chronic obstructive pulmonary disease
8. Subject who is pregnant.
9. Smoker (including ex-smoker and social smoker)
10. Chronic infective disease, including tuberculosis, hepatitis B and C; and HIV
11. Prior history of cancer (excludes pre-cancerous lesions)
12. Expected life expectancy less than 1 year
13. Known documented peripheral arterial disease
14. Known autoimmune disease or genetic disease
15. Known endocrine disease on treatment
16. Psychiatric illness
17. Previous stroke
18. Inability to comply with study protocol

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
No of participant with IL-11 detected in EBC and/or blood | 2 years
  A pilot study to optimize the feasibility of detection of IL-11 in EBC and blood, and other interleukins in blood of healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Chua Yang Chong, Principal Investigator, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Participants will be assigned a research ID that only research coordinator and team knows

REFERENCES:
- [Background] Serum interleukin-10 and interleukin-11 in patients in acute pancreatitis
- [Background] Ng B, Dong J, D'Agostino G, Viswanathan S, Widjaja AA, Lim WW, Ko NSJ, Tan J, Chothani SP, Huang B, Xie C, Pua CJ, Chacko AM, Guimaraes-Camboa N, Evans SM, Byrne AJ, Maher TM, Liang J, Jiang D, Noble PW, Schafer S, Cook SA. Interleukin-11 is a therapeutic target in idiopathic pulmonary fibrosis. Sci Transl Med. 2019 Sep 25;11(511):eaaw1237. doi: 10.1126/scitranslmed.aaw1237. PMID 31554736
- [Background] Ng B, Cook SA, Schafer S. Interleukin-11 signaling underlies fibrosis, parenchymal dysfunction, and chronic inflammation of the airway. Exp Mol Med. 2020 Dec;52(12):1871-1878. doi: 10.1038/s12276-020-00531-5. Epub 2020 Dec 1. PMID 33262481
- [Background] Ng B, Dong J, Viswanathan S, Widjaja AA, Paleja BS, Adami E, Ko NSJ, Wang M, Lim S, Tan J, Chothani SP, Albani S, Schafer S, Cook SA. Fibroblast-specific IL11 signaling drives chronic inflammation in murine fibrotic lung disease. FASEB J. 2020 Sep;34(9):11802-11815. doi: 10.1096/fj.202001045RR. Epub 2020 Jul 12. PMID 32656894
- [Background] Role of interleukins in the pathogenesis of pulmonary fibrosis
- [Background] Wu J, Chen J, Lv X, Yang Q, Yao S, Zhang D, Chen J. Clinical value of serum and exhaled breath condensate inflammatory factor IL-11 levels in non-small cell lung cancer: Clinical value of IL-11 in non-small cell lung cancer. Int J Biol Markers. 2021 Jun;36(2):64-76. doi: 10.1177/17246008211023515. Epub 2021 Jun 18. PMID 34142593
- [Background] She YX, Yu QY, Tang XX. Role of interleukins in the pathogenesis of pulmonary fibrosis. Cell Death Discov. 2021 Mar 15;7(1):52. doi: 10.1038/s41420-021-00437-9. PMID 33723241